CLINICAL TRIAL: NCT05087693
Title: Examining the Effect of Salbutamol Use in Asthma and/or Exercise Induced Bronchoconstriction Whilst Exercising in Ozone Air Pollution
Brief Title: Salbutamol Use in Ozone Air Pollution by People With Asthma and/or Exercise Induced Bronchoconstriction (EIB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Koehle, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H21-01080
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Asthma and/or Exercise Induced Bronchoconstriction; Ozone Air Pollution
Keywords: Asthma; Exercise Induced Bronchoconstriction; Salbutamol; Ozone
MeSH Terms: conditions — Asthma | interventions — Albuterol; Ozone; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Drug condition (placebo or salbutamol) will be double blinded Air quality condition (ozone or filtered air) will be single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Exercising in ozone following salbutamol inhalation (Experimental): Participants will be doing sub-maximal exercise (60% of VO2max for 30 minutes) on a cycle ergometer while inhaling 170ppb ozone after inhaling 200ug of salbutamol.
  Interventions: Drug: Salbutamol; Other: Ozone; Other: Exercise
- Exercising in filtered air following salbutamol inhalation (Active Comparator): Participants will be doing sub-maximal exercise (60% of VO2max for 30 minutes) on a cycle ergometer while inhaling filtered air after inhaling 200ug of salbutamol.
  Interventions: Drug: Salbutamol; Other: Filtered Air; Other: Exercise
- Exercising in ozone following placebo inhalation (Placebo Comparator): Participants will be doing sub-maximal exercise (60% of VO2max for 30 minutes) on a cycle ergometer while inhaling 170ppb ozone after inhaling placebo medication.
  Interventions: Drug: Placebo medication; Other: Ozone; Other: Exercise
- Exercising in filtered air following placebo inhalation (Placebo Comparator): Participants will be doing sub-maximal exercise (60% of VO2max for 30 minutes) on a cycle ergometer while inhaling filtered after inhaling placebo medication.
  Interventions: Drug: Placebo medication; Other: Filtered Air; Other: Exercise

INTERVENTIONS:
Drug: Salbutamol — Inhaling 200ug of salbutamol
  Arms: Exercising in filtered air following salbutamol inhalation; Exercising in ozone following salbutamol inhalation
Drug: Placebo medication — Inhaling placebo medication
  Arms: Exercising in filtered air following placebo inhalation; Exercising in ozone following placebo inhalation
Other: Ozone — Breathing 170ppb ozone
  Arms: Exercising in ozone following placebo inhalation; Exercising in ozone following salbutamol inhalation
Other: Filtered Air — Breathing filtered air
  Arms: Exercising in filtered air following placebo inhalation; Exercising in filtered air following salbutamol inhalation
Other: Exercise — Cycling at 60% of VO2max on a cycle ergometer

SUMMARY:
Salbutamol use is increased in areas with high levels of ozone pollution and the potential consequences of this are not well known. The purpose of this study is to examine the effect of salbutamol on lung function and inflammation in people with asthma and/or EIB exercising in ozone air pollution. To examine this, we are planning a randomized cross over trial where people with asthma and/or EIB complete sub maximal exercise in four conditions on four separate days. The four condition are: ozone + salbutamol, filtered air + salbutamol, ozone + placebo medication, and filtered air + placebo medication.

ELIGIBILITY:
Inclusion Criteria:

* Have asthma and/or EIB
* Able to perform maximal exercise
* Able to communicate sufficiently using the English language

Exclusion Criteria:

* Allergic to salbutamol (also known as Ventolin)
* Pregnant or potentially pregnant
* Have a history of smoking
* Had an upper respiratory tract infection within the last 4 weeks
* Have a chronic respiratory disease other than asthma or EIB

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Environmental Physiology Laboratory, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Any data shared will not contain any personal identifiers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Individuals without EIB were excluded. 23 tested positive for EIB, but only 18 were ultimately enrolled and scheduled for testing.
Groups:
- All Participants: Participants will be doing sub-maximal exercise (60% of VO2max for 30 minutes) on a cycle ergometer on four occasions in random order.
  On one of the occasions they will exercise while inhaling 170ppb ozone after inhaling 200ug of salbutamol.
  On one of the occasions they will exercise while inhaling 170ppb ozone after inhaling one puff of placebo.
  On one of the occasions they will exercise while room air after inhaling 200ug of salbutamol.
  On one of the occasions they will exercise while inhaling room air after inhaling one puff of placebo.
  Exercise: Cycling at 60% of VO2max on a cycle ergometer
  Due to the randomised nature there will be more than six possible sequences of these four exposures, thus as per guidance from clinical trials.gov we will use a single arm/group for the participant flow.
Period: Overall Study
Arm/Group | All Participants
Started | 18
Ozone/Placebo | 18
Ozone/Salbutamol | 18
Clean Air/Placebo | 18
Clean Air/Salbutamol | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants who screened positive and included in the 4 testing bouts.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 18

OUTCOME MEASURES:

1. Primary Outcome: Measured Before and 30 Minutes After Exercise in Each 1 Day Condition
Description: Measure of pulmonary function
Time Frame: Measured before and 30 minutes after exercise in each 1 day condition
Population: Entire study population
Measure: Mean (95% Confidence Interval); unit: litres
Arm/Group | Exercising in Ozone Following Salbutamol Inhalation | Exercising in Filtered Air Following Salbutamol Inhalation | Exercising in Ozone Following Placebo Inhalation | Exercising in Filtered Air Following Placebo Inhalation
Number analyzed (Participants) | 18 | 18 | 18 | 18
litres | 6.98 [5.25 to 8.71] | 5.96 [4.23 to 7.69] | -1.38 [-3.12 to .35] | -.35 [-2.08 to 1.39]

2. Primary Outcome: Change in FVC From Baseline to 30 Minutes After Exercise
Description: Measure of pulmonary function
Time Frame: Measured before and 30 minutes after exercise in each 1 day condition
Measure: Mean (95% Confidence Interval); unit: litres
Arm/Group | Exercising in Ozone Following Salbutamol Inhalation | Exercising in Filtered Air Following Salbutamol Inhalation | Exercising in Ozone Following Placebo Inhalation | Exercising in Filtered Air Following Placebo Inhalation
Number analyzed (Participants) | 18 | 18 | 18 | 18
litres | .77 [-.14 to 1.67] | .39 [-.51 to 1.29] | -1.37 [-2.28 to -.47] | -1.44 [-2.35 to -.54]

ADVERSE EVENTS:
Time Frame: Over the period from recruitment to completion of data collection for each individual. Five visits total over a period of approximately 10 days to 6 weeks.
Arm/Group | Exercising in Ozone Following Salbutamol Inhalation | Exercising in Filtered Air Following Salbutamol Inhalation | Exercising in Ozone Following Placebo Inhalation | Exercising in Filtered Air Following Placebo Inhalation
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT05087693/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT05087693/ICF_001.pdf